CLINICAL TRIAL: NCT00985478
Title: A Double-blind, Randomized, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SLV342 in Young Healthy Male Subjects
Brief Title: First in Man Study With SLV342
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated on 14 Sep 2010 due to strategic considerations
Sponsor: Abbott Products (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S342.1.001; 2009-014245-88 (EudraCT Number)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Pharmacokinetics
Keywords: First in Man; SLV342; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): SLV342 suspension or capsule
  Interventions: Drug: SLV342
- B (Placebo Comparator): matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SLV342 — 25 mg once daily - Maximal Tolerated Dose
  Arms: A
Drug: placebo — matching placebo
  Arms: B

SUMMARY:
First in man study with single and multiple rising doses with SLV342

ELIGIBILITY:
Inclusion Criteria

* Healthy

Exclusion Criteria

* Not healthy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters: adverse event, vital signs, 12-Lead ECG, continuous lead II ECG monitoring, laboratory safety variables and physical examination | 28 Days

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Plasma: Cmax, tmax, AUC, t½, λz, CL/F, and Vz/F. Urine: Aeurine, fe, and CLR | 28 days
Pharmacodynamic parameters: biochemistry and 24 h Holter monitoring | 28 days
Midazolam PK parameters | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Meuwsen, MS, Study Director — Abbott Healthcare Products B.V
Locations (1):
- Site Reference ID/Investigator# 61142, London, United Kingdom